CLINICAL TRIAL: NCT01477827
Title: Sunlight Exposure and Vitamin D Status of Children in the UK
Brief Title: Sunlight Exposure and Vitamin D in Children
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Lesley Rhodes, Professor of Experimental Dermatology, University of Manchester
Other Study IDs: Bupa Protocol 1
Record Dates: First submitted 2011-11-18; First posted 2011-11-23 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Schoolchildren

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy adolescents aged 12-15 years
  Interventions: Other: None - observational study

INTERVENTIONS:
Other: None - observational study

SUMMARY:
The purpose of this study is to examine the amount of sunlight exposure and vitamin D status of adolescent schoolchildren in each season throughout the year.

ELIGIBILITY:
Inclusion Criteria:

* Healthy school children aged 12-15 years
* White Caucasian
* Male or female

Exclusion Criteria:

* History of photosensitivity disorder

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Schoolchildren in Greater Manchester
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Serum concentration of 25-hydroxyvitamin D | Approximately every 3 months

SECONDARY OUTCOMES:
Amount of sunlight exposure received | Approx every 3 months
  Exposure to sunlight over 7 consecutive days is measured using polysulphone badges with one badge for weekdays and a second badge for the weekend.
Dietary intake of vitamin D | Approximately every 3 months
  Intake of foods containing vitamin D is recorded for a one week period and the average daily intake determined.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Rhodes, MBBS MD FRCP, Principal Investigator — University of Manchester
Locations (1):
- Salford Royal NHS Foundation Trust, Manchester, United Kingdom